CLINICAL TRIAL: NCT04113031
Title: Flywheel Squats Versus Free Weight High Load Squats for Explosive Actions in Football
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019/374030
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: SOCCER
Keywords: Sprint; Jump; Maximal Strength; Power

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Flywheel group (Experimental): The players allocated to the flywheel group will perform six weeks of squat resistance exercise using a flywheel device.
  Interventions: Behavioral: Flywheel squats versus free weight high load squats for explosive actions in football
- Barbell free weight group (Experimental): The players allocated to the barbell free weight group will perform six weeks of squat resistance exercise using a an olympic barbell and free weight of high loads.
  Interventions: Behavioral: Flywheel squats versus free weight high load squats for explosive actions in football
- Control (Active Comparator): All players in all three groups (including control group) will be instructed to adhere to their two-three weekly football practices and preseason matches of their team (~one weekly match).
  Interventions: Behavioral: Flywheel squats versus free weight high load squats for explosive actions in football

INTERVENTIONS:
Behavioral: Flywheel squats versus free weight high load squats for explosive actions in football — Over the course of the interventions, all players in all three groups will be instructed to adhere to their two-three weekly football practices and preseason matches of their team (~one weekly match). The flywheel group performes squat resistance exercise in using a flywheel device, and the barbell free weight group performes squat resistance exercise using an Olympic barbell and weights.

SUMMARY:
The objective of this randomized controlled trial is to compare the effect of flywheel resistance exercise versus free weight high load low velocity resistance exercise, where both modalities are carried out in a squat exercise with maximal intended mobilization of force contractions and combined with football practices, on 10 meter sprint, countermovement jump (CMJ) and one repeition maximum (1RM) partial 90° range of motion (ROM) squat strength in football players. The investigators 1) hypothesize that resistance exercise using flywheels and barbell free weights (BFW) combined with football practices will equally improve sprint time and jump height, and 2) the investigators hypothesize that squats carried out in a BFW exercise will result in superior improvements in 1RM partial squat compared with flywheel squats.

DETAILED DESCRIPTION:
The investigators will aim at recruiting 45 recreationally active football players, that will be randomly allocated to three groups: 1) flywheel (FW) group (n=15), 2) barbell free weight (BFW) group (n=15) and 3) control group (n=15).The FW and the BFW group will participate in an intervention where they perform a squat exercise either with a FW device or with BFWs twice a week over six weeks (in total 12 sessions) as a part of their preseason preparations. The control group will be instructed to not perform lower body resistance exercise and only to perform their teams' preseason preparations and acted as controls. During the intervention period, all players in all groups will be instructed to avoid other resistance exercises for their lower body, while no restrictions will be given in regard to resistance exercises for their upper body in their spare time.

This study will be carried out in accordance with international ethical standards for sport and exercise science and to the Declaration of Helsinki; prior to pre-tests, all the players will be informed of the purpose of the study and its associated risks and benefits, before providing oral and written informed consent. The Norwegian Data Protection Service has approved the study and the storage of personal data (Approval reference number: 374030). No further Regional Ethical approval per applicable institutional and national guidelines for sport and exercise science.

Prior to the interventions, the players will undergo pre-tests in the following order on the same test day: 1) 10 meter sprint time, 2) CMJ and 3) 1RM in a free barbell partial squat, carried out as 90° ROM in the knee joint (standing position = 180°).

10 meter sprint: The 10 meter sprint test will be performed on artificial grass indoors. Photocells mounted to the floor and walls recorded the sprint times, where the photocells at the starting and the finishing line are placed 20 cm and 100 cm above the ground, respectively. A marker is placed 30 cm behind of the starting timing gate, where the players chose their starting position behind the marker. The players starts their test on their own initiative, and without verbal encouragement, by breaking the laser beam at the starting timing gate and sprinted to the finishing line as fast as they can. Each player is given three attempts with three minutes recovery between each sprint.

Countermovement jump:

the players will test their jump height with a countermovement jump on a force platform that measures the vertical jump height in centimetres (cm) by calculating the centre of mass displacement from force development (take-off velocity) and body mass. Starting from an upright standing position with their feet shoulder-width apart and with both hands placed on their hips, the players will make a preliminary downward movement (eccentric phase) by flexing their hips and knees to approximately 90° (knee-flexion) before performing the concentric phase of the vertical jump off the ground by extending the knees and the hips, respectively. Each player is given three attempts with three minutes recovery between each jump.

One repetition maximum in squat:

Following the jump test, the players will perform a one repetition maximum (1RM) partial range of motion (90° knee joint angle) back squat test using an Olympic barbell. The players will warm up by lifting the Olympic barbell (20 kg) without additional weights for 8-10 repetitions, and thereafter perform two sets of progressively decreasing repetitions (6 and 3 repetitions, respectively) and increasing the weights based on their perceived effort in the previous warmup set. Thereafter, the players attempts their 1RM trials with increasing weights (2.5-10 kg) until failure. Failure is defined as inability to lift the barbell to standing (starting) position (180° knee joint angle). A goniometer will be held to the lateral part of their knee joint by an instructor to ensure that the players reach 90° of knee flexion before they are given a verbal "go" and they can start the concentric phase of the lift. The kilograms (kg) lifted in the last approved set is considered their 1RM and recorded in kg.

Exercise interventions Over the course of the interventions, all players in all three groups will be instructed to adhere to their two-three weekly football practices and preseason matches of their team (~one weekly match). The players in the FW and BFW groups start their exercise interventions the week following pre-tests. All intervention sessions were performed in the same laboratory and supervised by the same instructor. The players in both intervention groups are expected to experience a large increase in 1RM partial squat strength and thus a predominant increase in quadriceps muscle force is expectable with respects to hamstrings force. Therefore, the players will also perform the Nordic hamstring exercise to avoid a large quadriceps-to-hamstring strength ratio and thereby potentially reduce the risk for hamstring strains.The Nordic hamstring exercise will be performed at the end of each exercise session (for both interventions) and involve three sets of four repetitions (week 1) where the number of repetitions is progressively increasing to five in week 2, six in week 3-4, eight in week 5, and 10 in the final week of the interventions.

Flywheel group:

The players allocated to the FW group will be equipped with a west around their upper body connected with a band to the FW device (#215 YoYo Squat Unlimited Pro, nHance, YOYO Technology, Stockholm, Sweden). The players start in a deep squat position (~120° knee angle), and perform at first a standardized warmup set with six repetitions using the #1 inertia FW (0.025 kg·m-2). Thereafter, the players perform their maximal intended mobilization of force contraction sets by starting with three slow repetitions to allow the players to get into the flow of the squat exercise movement, where they will be given a verbal "go" when starting to push with maximal intended mobilization of force from deep squat starting position to standing position. The band connecting the west and the FW device will be strapped tightly making the players stop at 175° knee joint angle in the standing position when the FW band is unwound. When the FW continues to rewind again and produces kinetic force in the pivoting shaft, this immediately will force the players to bend their knees and begin the eccentric contraction phase. The players are instructed to over-win the kinetic energy with the highest possible mobilization of muscular force, and immediately start a new concentric maximal intended mobilization of force contraction. During the sets and sessions, the load (Watt) is monitored using the manufacturer´s application (Bluebrain, Kuopio, Finland) on a portable tablet (Samsung Galaxy S4, Samsung Electronics, Daegu, South Korea) connected to the FW device through Bluetooth. If the players produces on average >4 watts·kg-1 from each repetition of one set, the FW size is increased, to #2 (0.05 kg·m-2) and later to #3 (#1 + #2= 0.075 kg·m-2) and finally #4 (0.1 kg·m-2). Throughout the sessions, the players are given verbal encouragement. In week 1 and 2 of the intervention, the players will perform six sets with six repetitions, thereafter, in week 3, 4 and 5-6, the players will perform 3x5, 4x5 repetitions and 4x4 repetitions, respectively. Recovery time between sets is set to ≥3 minutes.

Barbell free weight sqaut group The BFW group performes a specialized warmup with three sets of progressively increasing intensity in the squat exercise; eight repetitions at 30%-, six repetitions at 50%- and six repetitions at 70% of 1RM, respectively. In all sessions, the players are instructed to perform the concentric phased lift with maximal intended mobilization of force and are given verbal encouragement throughout the sessions. The first two sessions (week 1) consists of familiarization to the squat exercise movement with three sets of eight repetitions at ~70% of 1RM. Thereafter, from the third session (week 2), the players are instructed to perform four sets of four repetitions with high loads (preferably >85% of 1RM) throughout the remaining sessions with progressively increasing the load with 5kg if they can perform five repetitions within one set.

ELIGIBILITY:
Inclusion Criteria:

* play at a adult (>16 years in Norway) football team that has an overall exercise load of two and/or three football practices in addition to one preseason football match a week.

Exclusion Criteria:

* Injuries that makes resistance exercise unachievable

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
10 meter sprint time | from baseline (pre-test) at week 1, to post-test, following six weeks of squat resistance exercise at week 7..
  change in seconds in 10 meter sprint time

SECONDARY OUTCOMES:
countermovement jump height | from baseline (pre-test) at week 1, to post-test, following six weeks of squat resistance exercise at week 7.
  change in centimeters jumped in countermovement jump height
one repetition maximum partial range of motion squat | from baseline (pre-test) at week 1, to post-test, following six weeks of squat resistance exercise at week 7.
  change in kilograms lifted in one repetition maximum partial range of motion squat
Weight | from baseline (pre-test) at week 1, to post-test, following six weeks of squat resistance exercise at week 7.
  change in kilograms measured as body mass

CONTACTS AND LOCATIONS:
Overall Officials: Svein Arne Pettersen, MSc, Principal Investigator — UiT The Arctic University of Norway
Locations (1):
- Lars Petter Rotvold Nilsen, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: No
Lars Petter R Nilsen and Edvard H Sagelv are the only two researchers with access to the data.

REFERENCES:
- [Derived] Sagelv EH, Pedersen S, Nilsen LPR, Casolo A, Welde B, Randers MB, Pettersen SA. Flywheel squats versus free weight high load squats for improving high velocity movements in football. A randomized controlled trial. BMC Sports Sci Med Rehabil. 2020 Oct 2;12:61. doi: 10.1186/s13102-020-00210-y. eCollection 2020. PMID 33024564